CLINICAL TRIAL: NCT04105985
Title: Kovanaze Vs. Articaine in Achieving Pulpal Anesthesia of Maxillary Teeth: A Randomized Clinical Trial
Brief Title: Kovanaze Vs. Articaine in Achieving Pulpal Anesthesia of Maxillary Teeth - Endodontics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer discontinued drug before any participants could be enrolled.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20014136 - adult endodontics
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Caries,Dental; Apical Periodontitis
Keywords: Necrotic teeth, root canals
MeSH Terms: conditions — Dental Caries; Periapical Periodontitis | interventions — Tetracaine; Oxymetazoline; Carticaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kovanaze Nasal Spray (endodontics) (Experimental): Adults (>18 years) who require non-surgical root canal treatment in maxillary anterior teeth
  Interventions: Drug: Kovanaze Nasal Spray
- Articaine Injections (endodontics) (Active Comparator): Adults (>18 years) who require non-surgical root canal treatment in maxillary anterior teeth
  Interventions: Drug: Articaine Injection

INTERVENTIONS:
Drug: Kovanaze Nasal Spray — Intra-nasal local anesthetic
  Other Names: Tetracaine HCl, Oxymetazoline HCl, NDC # 69803-100-10
  Arms: Kovanaze Nasal Spray (endodontics)
Drug: Articaine Injection — Local anesthetic
  Other Names: Septocaine
  Arms: Articaine Injections (endodontics)

SUMMARY:
The primary goal of the study is to compare the success rates of pulpal anesthesia (defined as ability to complete the intended dental procedure without the need for rescue anesthesia) between Kovanaze nasal mist and Articaine needle anesthesia.

DETAILED DESCRIPTION:
In June 2016, an intranasal delivery system of local anesthesia called Kovanaze, gained FDA approval. [9] Kovanaze is available as a 0.2 ml metered spray and is intended to achieve pulpal anesthesia of 5 maxillary teeth on either side of the face.

With the ability to avoid the traditional painful injection Kovanaze offers promise in the field of maxillary anesthesia and this study intends to:

1. Compare Kovanaze to conventional needle anesthetic for procedures other than fillings and/or involving multiple teeth in adults
2. Evaluate patient anxiety, tolerance and acceptability of Kovanaze in patients undergoing dental procedures

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Class I or II
* Preoperative heart rate of 55 to 100 beats per minute
* Maximum blood pressure reading of 166/100 mmHg
* Treatment for a pathology in the maxillary anterior tooth or premolar that requires administering local anesthesia
* Adults (>18 years) who require non-surgical root canal treatment in maxillary anterior teeth

Exclusion Criteria:

* Inadequately controlled thyroid disease
* Five or more nosebleeds in the past month
* Known allergy to any study drug or para-aminobenzoic acid
* History of methemoglobinemia
* Taking monoamine oxidase inhibitors, tricyclic antidepressants (i.e. amitriptyline), or non-selective beta adrenergic antagonists (i.e. propranolol);
* Taking oxymetazoline-containing products (i.e., Afrin) in the last 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Success rate of pupal anesthesia | immediately after dental procedure, an average of 3 hours
  % dental procedures completed without the need for rescue anesthesia

SECONDARY OUTCOMES:
Spread of anesthesia | immediately after dental procedure, an average of 3 hours
  Number of teeth anesthetized in maxillary arch
Change in Anxiety level | from baseline to immediately after dental procedure
  Modified Dental Anxiety Scale - 5 item questionnaire assessing dental visit related anxiety on a 5 point scale ranging from 1 (not anxious) to 5 (extremely anxious). Scores range from 5 to 25.
Change in Blood pressure | from baseline to immediately after dental procedure
Change in heart rate | from baseline to immediately after dental procedure
Change in pain | from baseline to immediately after dental procedure
  Heft-Parker visual analog scale rated from none (0mm) to maximum possible (170mm)
Satisfaction with Kovanaze | immediately after dental procedure, an average of 3 hours
  8-item questionnaire with a variety of scales designed to measure satisfaction with Kovanaze
Number of post treatment anesthesia side effects | 24 hours
  Phone survey asking about any side effects experienced from the anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Parthasarathy Madurantakam, DDS, PhD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No